CLINICAL TRIAL: NCT01104012
Title: The VAPARA Study: Validation of Proteomic Analyses for Allergic Asthma and Rhinitis
Brief Title: Validation of Proteomic Analyses for Allergic Asthma and Rhinitis
Acronym: VAPARA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2009/NM-01; 2009-A00399-48 (Other: Agence Française de Sécurité Sanitaire des Produits de Santé (Afssaps), RCB Number)
Record Dates: First submitted 2010-04-08; First posted 2010-04-15 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Rhinitis, Allergic; Asthma, Allergic
MeSH Terms: conditions — Rhinitis, Allergic; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma samples are taken on patient inclusion. For the purposes of this study, only proteomic profiles via SELDI-TOF will be characterized. Excess serum and plasma will be stored in the CHU de Nîmes Biothèque.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Allergy patients, asthma and rhinitis
  Interventions: Biological: Classification as "asthmatic" or "rhinitis only" via proteomic analysis; Biological: Classification as "asthmatic" or "rhinitis only" according to a metacholine test

INTERVENTIONS:
Biological: Classification as "asthmatic" or "rhinitis only" via proteomic analysis — Proteomic profiles are established for each patient using plasma and serum samples
Biological: Classification as "asthmatic" or "rhinitis only" according to a metacholine test — A positive metacholine test indicating bronchial hyperresponsiveness is currently our Gold Standard for diagnosing asthma.

SUMMARY:
The purpose of this study is to verify and validate the intrinsic diagnostic value in terms of sensitivity and specificity of proteomic profiles determined during a pre-study for discriminating between allergy related asthma and allergy related rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* signed consent
* never-smokers or non-smoking for at least 2 years + < 5 packs per year
* capable of understanding the study
* patient is affiliated with a social security system
* positive skin tests (at least one for Montpellier region pneumoallergens)
* treated with nasal or inhaled corticoids, leucotriene receptor antagonists, anti-IgE, Theophylline, anti-histamines, sodium cromoglycate, beta-blockers, benzodiazépine, oral corticoids: all these treatments must be interrupted for at least 72 hours

Exclusion Criteria:

* Co-morbidities: none; no co-morbidities are accepted
* dental infections (any) during the 3 months preceding the study
* suspected alcoholism or drug abuse
* chronic viral infection (hepatitis, HIV)
* patient under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The asthma and allergic rhinitis patients included in this study are recruted from the Pneumology Departments of the University Hospitals of Nîmes, Marseilles, and Montpellier.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Proteomic profile of each patient | One day (snapshot)
  The attribution of a proteomic profile as either "asthmatic" or "rhinitis". Proteomic profiles are determined accordig to the SELDI-TOF method. This is a transversal study validating proteomic profiles as a new diagnostic test.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Molinari, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - Assistance Publique - Hopitaux de Marseille, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nîmes, Nîmes